CLINICAL TRIAL: NCT01688479
Title: Randomized, Blinded Phase III Trial Comparing Calendula Officinalis Cream With Standard Aqueous Cream "Essex" for Treatment of Skin Reactions Caused by Postoperative Radiotherapy of Breast Cancer
Brief Title: Trial Comparing Calendula Officinalis With Aqueous Cream "Essex" to Treat Skin Reactions From Radiotherapy of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Hatschek, MD, PhD, Assoc. prof., Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Calendula trial
Record Dates: First submitted 2012-09-15; First posted 2012-09-20 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Postoperative Radiotherapy Breast Cancer
Keywords: Postoperative radiotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lanolin; Sesame Oil; Parabens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calendula Weleda® cream (Weleda) (Experimental): Calendula Officinalis (marigold plant) is applied twice daily on the skin in the radiated area during the entire treatment period and until the skin reaction subsided
  Interventions: Drug: Calendula Weleda cream (Weleda AG, Sweden) contains extracts of marigold plant (Calendula Officinalis 10%), wool fat and sesame oil
- Essex® cream (Schering-Plough) (Active Comparator): Essex cream is applied twice daily on the skin in the radiated area during the entire treatment period and until the skin reaction subsided
  Interventions: Drug: Essex® cream (Schering-Plough), aqueous cream without parabens

INTERVENTIONS:
Drug: Calendula Weleda cream (Weleda AG, Sweden) contains extracts of marigold plant (Calendula Officinalis 10%), wool fat and sesame oil
  Arms: Calendula Weleda® cream (Weleda)
Drug: Essex® cream (Schering-Plough), aqueous cream without parabens
  Arms: Essex® cream (Schering-Plough)

SUMMARY:
Acute radiation skin reactions (ARSR) occur in the majority of patients undergoing postoperative radiotherapy (RT). Some patients experience more severe reactions such as dry and/or moist desquamation but most patients experience mild reactions e.g. erythema (Lopez et al., 2005). The radiation dose, volume, RT technique and previous treatment, such as type of surgery and previous chemotherapy, are factors that might impact on the risk for ARSR together with patient-related factors such as body mass index (BMI), smoking status and previous skin damage (Porock et al., 1998; Wells et al., 2004). In a pilot study (n=93) of the frequency of ARSR in patients with breast cancer who underwent adjuvant RT it was shown that 93% developed ARSR, mostly mild reactions. Patients reported low scores on pain and itching (Sharp et al., 2011). Over 80% of the patients reported adherence to the skin care recommendations which included application of a thin layer of Essex® cream, a non-perfumed aqueous cream, on the irradiated area at least two times a day (Sharp et al., 2011). The effects of skin care products containing Calendula Officinalis (marigold plant) on ARSR in patients with breast cancer were investigated in a randomized clinical trial (Pommier et al., 2004). Patients in the experimental group, treated with calendula cream had a statistically significant lower incidence of severe ARSR, pain and treatment interruptions in comparison with the patients in the control group, treated with trolamine.

The purpose of this blinded, randomized clinical trial is to compare two topical agents, Calendula Weleda® cream and Essex® cream, in terms of efficacy to reduce the risk of severe acute radiation skin reactions (ARSR) in relation to adjuvant radiotherapy (RT) for breast cancer.

Patients were instructed to apply a thin layer of the assigned cream twice a day, starting at the onset of RT and continue until two weeks after termination, or until the ARSR is healed. The application should include the whole treatment area including the armpit and shoulder/back area in patients treated with modified radical mastectomy. Patients are also advised to not apply the cream within two hours before the RT in order to avoid possible build-up effect. Daily wash with perfume free soap and tap water are recommended and patients are advised to refrain from use of other topical agents in the irradiated area.

The primary endpoint is the efficacy to reduce acute radiation skin reactions (ARSR), assessed with the Radiation Therapy Oncology Group/The Organization for Research and Treatment of Cancer Acute Radiation Morbidity Scoring Criteria (RTOG/EORTC scale) at follow-up.

Secondary endpoints include patient reported outcome measures; Quality of Life Questionnaire (QLQ-C30), Sleep disturbances (MOS-sleep questionnaire) and symptoms experienced from the irradiated area (visual analogue scale). Patients' experiences and adherence to the topical agents are also evaluated.

A total of 400 patients are required to detect a true absolute reduction in the proportion of patients with ARSR, from 35% with standard treatment (Essex® cream) to 20% with the experimental treatment (Calendula Weleda® cream), with a significance level of 5% a power of 90%. With this sample size, 95% confidence intervals for the difference in proportions are estimated to be in the order of ±10%. Assuming a rate of 5% of non-responders, the target size has been set to 420 patients.

ELIGIBILITY:
Inclusion Criteria:

* radically operated for breast cancer,
* aged 18 years or older,
* signed informed consent

Exclusion Criteria:

* previous radiation in the same area,
* severe general health problems,
* ECOG performance status > 3,
* reduced cognitive ability,
* allergy to marigold plant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Grade of skin reactions to radiotherapy | 8 weeks
  Skin reactions due to radiotherapy using RTOG scale

SECONDARY OUTCOMES:
Quality of life in relation to skin reaction | 8 weeks
  Measurements of sleep disturbances acc. to the MOS-SLEEP scale and QoL acc. to EORTC QLQ-C30

OTHER OUTCOMES:
Impact of smoking habits on the intensity of the skin reaction | 8 weeks
  Collection of data on smoking habits and measurements of carbon monoxide in exhaled air

CONTACTS AND LOCATIONS:
Overall Officials: Maria AC Bergenmar, PhD, Principal Investigator — Dept of Oncology, Karolinska University Hospital, Stockholm, Sweden; Lena Sharp, PhD, Principal Investigator — Dept of Oncology, Karolinska University Hospital, Stockholm, Sweden; Thomas Hatschek, MD, PhD, Study Chair — Dept of Oncology, Karolinska University Hospital, Stockholm, Sweden
Locations (1):
- Department of Oncology, Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Result] Sharp L, Finnila K, Johansson H, Abrahamsson M, Hatschek T, Bergenmar M. No differences between Calendula cream and aqueous cream in the prevention of acute radiation skin reactions--results from a randomised blinded trial. Eur J Oncol Nurs. 2013 Aug;17(4):429-35. doi: 10.1016/j.ejon.2012.11.003. Epub 2012 Dec 13. PMID 23245940
- [Result] Sharp L, Johansson H, Hatschek T, Bergenmar M. Smoking as an independent risk factor for severe skin reactions due to adjuvant radiotherapy for breast cancer. Breast. 2013 Oct;22(5):634-8. doi: 10.1016/j.breast.2013.07.047. Epub 2013 Aug 13. PMID 23953136